CLINICAL TRIAL: NCT00867451
Title: A Pilot Study Designed To Improve Sleep and Subsequent Daytime Functioning in Children Diagnosed With ADHD
Brief Title: Improving Sleep and Daytime Functioning Among Children Diagnosed With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHMC IRB# 2008-1287
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Treatment (Experimental): Children will receive behavioral sleep interventions and, if needed, melatonin, to improve sleep functions.
  Interventions: Behavioral: Sleep Intervention; Drug: Melatonin
- Delayed Treatment (Experimental): Children will only receive sleep behavior interventions for the first four weeks of the trial. Treatment with study drug will be delayed to the 5th week.
  Interventions: Behavioral: Sleep Intervention; Drug: Melatonin

INTERVENTIONS:
Behavioral: Sleep Intervention — A structured sleep protocol is taught to parents, use of a white noise generator
Drug: Melatonin — Body Weight <40mg will be given 3mg at bedtime for two weeks Body Weight >40mg will be given 6 mg at bedtime for two weeks

SUMMARY:
This study will test the efficacy of a systematic, multi-modal intervention protocol designed to improve sleep functioning and subsequent alleviation of daytime cognitive and behavioral difficulties among children diagnosed with ADHD. It is hypothesized that children receiving behavioral and (if necessary) pharmacologic interventions targeting sleep will display improvement on objective and subjective sleep measures, neuropsychological tests, and teacher-, and parent-ratings of ADHD behaviors.

DETAILED DESCRIPTION:
Parents, researchers, and clinicians have long suspected that inadequate sleep in many children diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) can exacerbate symptoms of hyperactivity and inattentiveness, leading to further cognitive and behavioral disruptions. Extant sleep studies report that upwards of 50% of children diagnosed with ADHD display behaviors associated with chronic sleep disruption (in comparison to non-diagnosed youth). Although studies have attempted to alleviate sleep difficulties, most intervention studies have used only one treatment modality. This study will incorporate a systematic, multi-method treatment intervention protocol that will combine behavioral and pharmacologic strategies aimed to improve sleep functioning among children with ADHD.

The specific aims of this study are to (a) examine the effects of a structured sleep behavioral/pharmacologic intervention protocol on improved sleep onset and efficiency, and (b) examine how such improvements may alleviate daytime neuropsychological (i.e., response time) and behavioral deficits associated with ADHD. The study will take place at the ADHD Clinic. Twelve children (ages 6-12), following confirmed diagnosis of ADHD and who meet all criteria for evaluation, and who have signed parent/child consent/assent, will be randomly assigned to an immediate treatment or delayed treatment group (6 in each group). Children in the immediate treatment group will receive the sleep intervention protocol, while those in the delayed treatment group will initially only receive all of the sleep, activity, and daytime assessments on the same schedule as the treatment group without any of the treatment methods. They will be offered the same treatment methods as the immediate treatment group at week 5.

The study will occur in separate phases. Phase one will consist of an intake session at the ADHD Clinic to determine eligibility for the study. Phase two will immediately follow (for eligible participants) and will consist of a one-week baseline to gather sleep, neuropsychological functioning and daytime behavior data. Sleep functioning will be measured using both subjective (i.e., parent sleep logs) and objective measures (i.e., actigraphy), while response time will be assessed using a device that measures continuous reaction-time performance. Attention and other ADHD-related behaviors will be collected using parent- and teacher rating scales during baseline. Phase three, which will last 4 weeks, consists of parents of each child in the treatment group coming to the Clinic to learn a specific sequence of interventions, first beginning with behavioral methods, followed by melatonin (if necessary) to improve sleep functioning (80% above baseline). Parents of children in the delayed treatment phase will not come to the Clinic during phase three, but will be contacted for a brief phone interview once per week. They will be asked questions pertaining to any changes in sleep and daytime behaviors. Finally, Phase 4 consists of having all parents return to the ADHD Clinic, where measures administered at the end of Baseline will be repeated. At that time, those in the delayed treatment group may enter the treatment phase. A repeated measure ANOVA using group status (no treatment vs. treatment) across two time points (baseline, post-sleep intervention) will assess changes in sleep and daytime functioning over time. Although a group-by-time interaction will indicate treatment efficacy, this is a small pilot study; the small number of participants in each group likely precludes the power to determine this statistically. Instead, effect sizes and subjective measures will be used to describe and justify, if appropriate, an expansion of this study for a subsequent grant application.

ELIGIBILITY:
Inclusion Criteria:

* Consent: The family must provide signature of informed consent by parents or legal guardians
* Assent: Children must provide assent to participate in the study (via signature on assent form)
* Age at time of Screening: 6 years to 12 years, inclusive
* Gender: includes male and female children.
* ADHD Diagnostic Status: The primary criterion is that patients must meet DSM-IV criteria for ADHD.
* Presence of Significant Sleep Problems: Assessed through clinical history and a commonly used parent-report of children's sleep habits. A cut-off score of or greater than 41 on the Children's Sleep Habits Questionnaire (CSHQ) will be used.
* Functioning at appropriate grade level for age.

Exclusion Criteria:

* Understanding Level: The parent is not fluent in the language of the wording used in the consent form.
* Exclusionary Psychiatric Conditions or Current Significant Stressors: Children whose primary diagnosis is something other than ADHD will be excluded from participation (e.g., oppositional defiant disorder, anxiety). Further, events that have occurred over the past 6 months that could affect sleep (such as active grieving) will also be excluded from participation.
* Developmental Disabilities: Functioning below grade level for age; or as a result of scores on the IQ screening, additional assessments, or the judgment of the study clinicians, patients will be excluded if they are deemed to be significantly developmentally delayed. This includes clinically significant delays in cognitive function or the presence of other Pervasive Developmental Disorders (PDD).
* Organic Brain Injury: Children must not have a history of head trauma (requiring hospitalization), neurological disorder (such as Tourette syndrome, or restless leg movements), or any other organic disorder that could possibly affect brain function.
* Strong evidence of sleep apnea: As determined by cutoff scores on the sleep habits questionnaire. Raw scores of or greater than 6 on relevant items from the CHSQ are often used to indicate sleep apnea.
* Caffeine consumption: is greater than 3 cans per day
* Stimulant or psychotropic medications: Children must be on a stable dose one week prior to the initiation of the study interventions and not require changes or addition of new medication during the intervention time.
* ADHD Medications:Children must be on a stable dose one week prior to the initiation of the study interventions and not require changes or addition of new medication during the intervention time.
* Child-bearing potential: Female subjects who are randomized to the treatment group and who are potentially able to become pregnant, must be willing to take adequate precautions to prevent pregnancy, as determined by the investigator.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gilman, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the community and families seeking services at the ADHD Clinic and in the Division of Developmental and Behavioral Pediatrics at Cincinnati Childrens Hospital Medical Center.
Groups:
- Immediate Treatment: Children immediately received behavioral sleep interventions (following a structured pre-bedtime routine protocol, incorporating a white noise machine during sleep) for two weeks. If sleep parameters did improve (80% from baseline), melatonin (3mg, administered orally 1 hour prior to bedtime) supplemented the behavioral sleep treatments, for two weeks. None of the participants improved their sleep by 80% from baseline using the behavioral treatments. Thus, all participants progressed to the melatonin phase of the intervention.
- Delayed Treatment: Pre-intervention data was collected for four weeks, after which children received behavioral sleep interventions (following a structured pre-bedtime routine protocol, incorporating a white noise machine during sleep) for two weeks. If sleep parameters did improve (80% from baseline), melatonin (3mg, administered orally 1 hour prior to bedtime) supplemented the behavioral sleep treatments, for two weeks. None of the participants improved their sleep by 80% from baseline using the behavioral treatments. Thus, all participants in the delayed treatment group progressed to the melatonin phase of the intervention.
Period: Overall Study
Arm/Group | Immediate Treatment | Delayed Treatment
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Delayed Treatment | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.3) | 9.5 (1.9) | 9.0 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Sleep Duration
Description: Data was gathered via actigraphy. Data was gathered on a nightly basis for one week at baseline and at week five. Data presented is the mean nightly value (in minutes) for that week.
Time Frame: Baseline; Week 5
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Baseline; Week 5: Results based on all participants (i.e., immediate and delayed-treatment participants).
Arm/Group | Baseline | Week 5
Number analyzed (Participants) | 8 | 8
minutes | 609.57 (25.54) | 602.79 (25.92)
Statistical Analysis 1: Comparison: Baseline; Test type: Superiority or Other; p < .05, t-test, 1 sided

2. Primary Outcome: Sleep Activity (i.e., Average Amount of Time That the Participant Moved During Sleep)
Description: Data was gathered via actigraphy. Data was gathered on a nightly basis for one week at baseline and at week five. Data presented is the mean nightly value (in minutes) of movement during sleep, for that respective week.
Time Frame: Baseline; Week 5
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Baseline | Week 5
Number analyzed (Participants) | 8 | 8
minutes | 31.25 (19.00) | 24.89 (11.72)

3. Primary Outcome: Length of Awake Time
Description: Data was gathered via actigraphy. Data was gathered on a nightly basis for one week at baseline and at week five. Data presented is the mean nightly value (in minutes) for that respective week.
Time Frame: Baseline; Week 5
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Baseline | Week 5
Number analyzed (Participants) | 8 | 8
minutes | 36.52 (20.20) | 19.81 (17.59)

4. Primary Outcome: Percent Total Sleep
Description: Data was gathered via actigraphy. Data on percentage of time individual was immobile during sleep was gathered on a nightly basis for one week at baseline and at week five. Data presented is the mean nightly percentage of immobility for that respective week.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: percentage of immobility
Arm/Group | Baseline | Week 5
Number analyzed (Participants) | 8 | 8
percentage of immobility | 82.02 (14.50) | 85.05 (12.50)

5. Primary Outcome: Vanderbilt ADHD Rating Scales - Teacher (VADTRS): Inattention
Description: 35-item measure to assess behaviors consistent with ADHD. Nine items reflected the Inattention scale. Range of scores for the Attention Problems domain was 0-27. Higher scores are indicative of higher levels of inattention.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Assessment; Week 5: Results based on all participants (i.e., immediate and delayed treatment participants).
Arm/Group | Baseline Assessment | Week 5
Number analyzed (Participants) | 8 | 8
units on a scale | 21.29 (3.03) | 18.00 (7.64)

6. Primary Outcome: Vanderbilt ADHD Rating Scales - Parent (VADPRS): Inattention
Description: as for outcome 5
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline Assessment | Week 5
Number analyzed (Participants) | 8 | 8
units on a scale | 21.29 (3.03) | 13.42 (6.45)

7. Primary Outcome: Vanderbilt ADHD Rating Scales - Teacher (VADTRS): Hyperactivity/Impulsivity
Description: 35-item measure to assess behaviors consistent with ADHD. Nine items reflected the Inattention scale. Range of scores for the Hyperactivity/Impulsivity domain was 0-27. Higher scores are indicative of higher levels of hyperactive/impulsive behaviors.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Assessment; Week 5: Results based on all participants (i.e., immediate and delays treatment participants).
Arm/Group | Baseline Assessment | Week 5
Number analyzed (Participants) | 8 | 8
units on a scale | 8.88 (7.31) | 7.50 (6.02)

8. Primary Outcome: Vanderbilt ADHD Rating Scales - Parent (VADPRS): Hyperactivity/Impulsivity
Description: as for outcome 7
Time Frame: Baseline, Week 35
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline Assessment | Week 5
Number analyzed (Participants) | 8 | 8
units on a scale | 15.29 (6.89) | 13.42 (6.42)

ADVERSE EVENTS:
Arm/Group | Immediate Treatment | Delayed Treatment
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes